CLINICAL TRIAL: NCT02821754
Title: A Pilot Study of Combined Immune Checkpoint Inhibition in Combination With Ablative Therapies in Subjects With Hepatocellular Carcinoma (HCC) or Biliary Tract Carcinomas (BTC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160135; 16-C-0135
Record Dates: First submitted 2016-06-29; First posted 2016-07-04 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Biliary Tract Neoplasms; Liver Cancer; Hepatocellular Carcinoma; Cholangiocarcinoma; Bile Duct Cancer
Keywords: PDL1-Mediated Adaptive Resistance; Monoclonal Antibody; CTLA-4; Ablative Therapy; Combination of Tremelimumab and Durvalumab
MeSH Terms: conditions — Biliary Tract Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma; Bile Duct Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — durvalumab; tremelimumab; Radiofrequency Ablation; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1/A1-Durvalumab + Tremelimumab (Experimental): Durvalumab + Tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- 2/A2 - Durvalumab + Tremelimumab + Trans-arterial Catheter Chemoembolization (TACE) (Experimental): Durvalumab + Tremelimumab + TACE
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Procedure: Trans-arterial Catheter Chemoembolization (TACE)
- 3/A3 - Durvalumab + Tremelimumab+ Radiofrequency Ablation (RFA) (Experimental): Durvalumab + Tremelimumab+ RFA
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Procedure: Radiofrequency Ablation (RFA)
- 4/A4 - Durvalumab + Tremelimumab+ Cryoablation (Experimental): Durvalumab + Tremelimumab+ Cryoablation
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Procedure: Cryoablation

INTERVENTIONS:
Drug: Durvalumab — Flat dose of 1500 mg every 4 weeks.
  Other Names: Imfinzi
Drug: Tremelimumab — Flat dose of 75 mg every 4 weeks for up to 4 doses.
  Other Names: Ticilimumab
Procedure: Trans-arterial Catheter Chemoembolization (TACE) — TACE will be performed on Day 36 (+/-96hrs).
  Other Names: TACE
  Arms: 2/A2 - Durvalumab + Tremelimumab + Trans-arterial Catheter Chemoembolization (TACE)
Procedure: Radiofrequency Ablation (RFA) — RFA will be performed on Day 36 (+/-96hrs).
  Other Names: RFA
  Arms: 3/A3 - Durvalumab + Tremelimumab+ Radiofrequency Ablation (RFA)
Procedure: Cryoablation — Cryoablation will be performed on Day 36 (+/-96hrs).
  Other Names: Cryosurgery
  Arms: 4/A4 - Durvalumab + Tremelimumab+ Cryoablation

SUMMARY:
BACKGROUND:

* Various tumor ablative procedures and techniques have been shown to result in immunogenic cell death and induction of a peripheral immune response. The term ablative therapies applies to trans-arterial catheter chemoembolization (TACE), radiofrequency ablation (RFA) and cryoablation (CA).
* The underlying hypothesis of this study is that the effect of immune checkpoint inhibition can be enhanced by TACE, CA and RFA in patients with advanced hepatocellular carcinoma (HCC) and biliary tract carcinomas (BTC). We have already demonstrated proof of principle as well as safety and feasibility of this approach with anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) therapy.
* Based on the concept of programmed death-ligand 1 (PDL1)-mediated adaptive resistance and the emerging role of programmed cell death protein 1 (PD1) therapy in HCC, we would like to evaluate the combination of tremelimumab and durvalumab (with ablative therapies) in HCC and BTC.

Objectives:

- To preliminarily evaluate the 6-month progression free survival (PFS) of combining tremelimumab and durvalumab in patients with advanced HCC (either alone or with cryoablation, TACE or RFA) and in patients with advanced biliary tract carcinoma (BTC) (either alone or with cryoablation or RFA).

ELIGIBILITY:

* Histologically or cytologically confirmed diagnosis of HCC or biliary tract carcinoma OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC (or biliary tract carcinoma).
* Childs-Pugh A/B7 cirrhosis only is allowed. If patient does not have cirrhosis, this limitation does not apply.
* Patients must have disease that is not amenable to potentially curative resection, radiofrequency ablation, or liver transplantation.

DESIGN:

We will evaluate the combination of tremelimumab and durvalumab (with ablative therapies) in cohorts A (HCC; N=40) and B (BTC; N=30). The first N=10 patients in both cohorts will receive tremelimumab and durvalumab only (i.e. No interventional radiologic procedures).

* A: Advanced HCC, BCLC# Stage B/C

  * N= 1st 10 pts: No ablative procedure Cryoablation/RFA/TACE##
  * Tremelimumab 75mg flat dose every (q)28 days for 4 doses; Durvalumab 1500mg flat dose q28 days until end of study (EOS)###
  * 40 total: 10 trem+ dur alone; 10 trem+ dur + TACE; 10 trem + dur + RFA; 10 trem + dur + cryo
* B: Intra/extra-hepatic cholangiocarcinoma

  * N= 1st 10 patients (pts): No ablative procedure; RFA/ cryoablation
  * Tremelimumab 75mg flat dose q28 days for 4 doses; Durvalumab 1500mg flat dose q28 days until EOS###
  * 30 total: 10 trem+ dur alone; 10 trem + dur + RFA; 10 trem

    * BCLC = Barcelona clinic liver cancer staging system

      * For BCLC stage B patients TACE may be repeated as per standard of care

        * EOS = End of study treatment or meeting any of the off-treatment or off study criteria.

DETAILED DESCRIPTION:
BACKGROUND:

* Various tumor ablative procedures and techniques have been shown to result in immunogenic cell death and induction of a peripheral immune response. The term ablative therapies applies to trans-arterial catheter chemoembolization (TACE), radiofrequency ablation (RFA) and cryoablation (CA).
* The underlying hypothesis of this study is that the effect of immune checkpoint inhibition can be enhanced by TACE, CA and RFA in patients with advanced hepatocellular carcinoma (HCC) and biliary tract carcinomas (BTC). We have already demonstrated proof of principle as well as safety and feasibility of this approach with anti-CTLA4 therapy.
* Based on the concept of PDL1-mediated adaptive resistance and the emerging role of PD1 therapy in HCC, we would like to evaluate the combination of tremelimumab and durvalumab (with ablative therapies) in HCC and BTC.

Objectives:

- To preliminarily evaluate the 6-month progression free survival (PFS) of combining tremelimumab and durvalumab in patients with advanced HCC (either alone or with cryoablation, TACE or RFA) and in patients with advanced biliary tract carcinoma (BTC) (either alone or with cryoablation or RFA).

ELIGIBILITY:

* Histologically or cytologically confirmed diagnosis of HCC or biliary tract carcinoma OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC (or biliary tract carcinoma).
* Childs-Pugh A/B7 cirrhosis only is allowed. If patient does not have cirrhosis, this limitation does not apply.
* Patients must have disease that is not amenable to potentially curative resection, radiofrequency ablation, or liver transplantation.

DESIGN:

We will evaluate the combination of tremelimumab and durvalumab (with ablative therapies) in cohorts A1 (HCC; Barcelona clinic liver cancer staging system (BCLC) stage C; N=10), A2 (HCC; BCLC stages B/C; N=30) and B (BTC; N=30). The patients in cohort A1 and first 10 patients in cohort B will receive tremelimumab and durvalumab only (i.e. no interventional radiologic procedures).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have histopathological confirmation of hepatocellular carcinoma (HCC) or biliary tract carcinoma (BTC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC (or biliary tract carcinoma). Fibrolamellar variant is also allowed. The term BTC includes intra or extrahepatic cholangiocarcinoma, gallbladder cancer or ampullary cancer.
  2. Patients must have disease that is not amenable to potentially curative resection, transplantation or ablation. HCC patients must have progressed on, been intolerant to, or refused prior sorafenib therapy. Patients with BTC must have received, been intolerant of or refused at least one line of chemotherapy.
  3. Patients must have multiple tumor lesions (at least 2): one for the ablation procedure and another for evaluation located outside the proposal ablation zone.
  4. Disease must be technically amenable to transhepatic arterial chemoembolization (TACE) (HCC patients only), radiofrequency ablation (RFA), or cryoablation. Each case will be discussed at gastrointestinal (GI) tumor board with interventional radiology. Patients must have evaluable disease.
  5. If liver cirrhosis is present, patient must have a Child-Pugh A/B7 classification
  6. Age 18 years or older
  7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
  8. Patients must have normal organ and marrow function as defined below:
* leukocytes greater than or equal to 3,000/mcL
* absolute neutrophil count greater than or equal to 1,000/mcL
* platelets greater than or equal to 60,000/mcL
* total bilirubin If cirrhosis present: Part of Child Pugh requirement; If no cirrhosis: bilirubin should be less than or equal to 2 x upper limit of normal (ULN)
* serum albumin If cirrhosis present: Part of Child Pugh requirement; If no cirrhosis: albumin should be less than or equal to 2.5g/dl
* patients are eligible with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) up to 5 x ULN.
* creatinine < 1.5x institution upper limit of normal OR creatinine clearance greater than or equal to 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal

  9. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.

  10. Patients must not have other invasive malignancies within the past 5 years (with the exception of non-melanoma skin cancers, non-invasive bladder cancer or localized prostate cancer for whom systemic therapy is not required).

  11. Patient must be able to understand and willing to sign a written informed consent document.

  12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women greater than or equal to 50 years of age would be considered post-menopausal if they have been

amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

13. Body weight greater than 30kg

EXCLUSION CRITERIA:

1. Patients who have had standard of care chemotherapy, large field radiotherapy, or major surgery must wait 2 weeks prior to entering the study. For recent experimental therapies a 28 day period of time must elapse before treatment.
2. Patients who have undergone prior liver transplantation are ineligible.
3. Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations that would limit compliance with study requirements.
5. History of chronic autoimmune disease (e.g., Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, rheumatoid arthritis, hypophysitis, etc.) with symptomatic disease within the 3 years before randomization. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion.
6. Dementia or significantly altered mental status that would prohibit the understanding or rendering of Information and Consent and compliance with the requirements of the protocol.
7. Diverticulitis either active or history of within the past 2 years. Note that diverticulosis is permitted.
8. Active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis. Currently receiving immunosuppressive doses of steroids or other immunosuppressive medications (inhaled and topical steroids are permitted)
9. History of sarcoidosis syndrome
10. Patients should not be vaccinated with live attenuated vaccines within 30 days of starting durvalumab or tremelimumab treatment.
11. Has a known history of Human Immunodeficiency Virus (HIV). HIV-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and tremelimumab. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that tremelimumab may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events.
12. History of hypersensitivity reaction to human or mouse antibody products.
13. Pregnancy and breast feeding are exclusion factors. The effects of tremelimumab on the developing human fetus are unknown. Enrolled patients must agree to use adequate contraception prior to study entry, the duration of study participation and 6 months after the end of the treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
14. Patients with unhealed surgical wounds for more than 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  In addition, all large scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
  Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Duffy AG, Greten TF. Immunological off-target effects of standard treatments in gastrointestinal cancers. Ann Oncol. 2014 Jan;25(1):24-32. doi: 10.1093/annonc/mdt349. Epub 2013 Nov 7. PMID 24201974
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Sangro B, Gomez-Martin C, de la Mata M, Inarrairaegui M, Garralda E, Barrera P, Riezu-Boj JI, Larrea E, Alfaro C, Sarobe P, Lasarte JJ, Perez-Gracia JL, Melero I, Prieto J. A clinical trial of CTLA-4 blockade with tremelimumab in patients with hepatocellular carcinoma and chronic hepatitis C. J Hepatol. 2013 Jul;59(1):81-8. doi: 10.1016/j.jhep.2013.02.022. Epub 2013 Mar 4. PMID 23466307
- [Derived] Myojin Y, Babaei S, Trehan R, Hoffman C, Kedei N, Ruf B, Benmebarek MR, Bauer KC, Huang P, Ma C, Monge C, Xie C, Hrones D, Duffy AG, Armstrong P, Kocheise L, Desmond F, Buchalter J, Galligan M, Cantwell C, Ryan R, McCann J, Bourke M, Mac Nicholas R, McDermott R, Awosika J, Cam M, Krebs R, Budhu A, Revsine M, Figg WD, Kleiner DE, Redd B, Wood BJ, Wang XW, Korangy F, Claassen M, Greten TF. Multiomics analysis of immune correlatives in hepatocellular carcinoma patients treated with tremelimumab plus durvalumab. Gut. 2025 May 7;74(6):983-995. doi: 10.1136/gutjnl-2024-334026. PMID 39965889
- [Derived] Monge C, Xie C, Myojin Y, Coffman-D'Annibale KL, Hrones D, Brar G, Wang S, Budhu A, Figg WD, Cam M, Finney R, Levy EB, Kleiner DE, Steinberg SM, Wang XW, Redd B, Wood BJ, Greten TF. Combined immune checkpoint inhibition with durvalumab and tremelimumab with and without radiofrequency ablation in patients with advanced biliary tract carcinoma. Cancer Med. 2024 Feb;13(3):e6912. doi: 10.1002/cam4.6912. Epub 2024 Jan 11. PMID 38205877
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0135.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled but not treated. With the exception of baseline data, no other data were collected for these participants.
Groups:
- Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE): RFA/TACE Tremelimumab (trem) 75mg flat dose every (q)28 days for 4 doses and Durvalumab (dur) 1500mg flat dose q28 days until end of study.
  30 total (e.g. Per the study design, this is the number of participants we planned to treat): 10 trem+ dur alone; 10 trem + dur + RFA; 10 trem + dur + cryoablation
- Radiofrequency Ablation/Cryoablation (RFA/CA): Tremelimumab (trem) 75mg flat dose every (q)28 days for 4 doses and Durvalumab (dur) 1500mg flat dose q28 days until end of study.
  30 total (e.g. Per the study design, this is the number of participants we planned to treat): 10 trem+ dur alone; 10 trem + dur + RFA; 10 trem + dur + cryoablation
- Enrolled But Not Treated: Enrolled but not treated.
Period: Overall Study
Arm/Group | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) | Radiofrequency Ablation/Cryoablation (RFA/CA) | Enrolled But Not Treated
Started | 36 | 16 | 2 (No results data were collected for these participants.)
Completed | 20 | 4 | 0
Not Completed | 16 | 12 | 2
Not completed — Procedure not required prior to amendment change | 13 | 11 | 0
Not completed — Participant's Clinical status | 2 | 0 | 0
Not completed — Participant removed for noncompliance | 1 | 0 | 0
Not completed — Drug not available. | 0 | 0 | 1
Not completed — Participant declined to participate (before treatment started.) | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) | Radiofrequency Ablation/Cryoablation (RFA/CA) | Enrolled But Not Treated | Total
Number analyzed (Participants) | 36 | 16 | 2 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 12 | 1 | 30
  >=65 years | 19 | 4 | 1 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.54 (12.57) | 57.59 (14.24) | 66.1 (3.25) | 62.54 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 1 | 16
  Male | 27 | 10 | 1 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 0 | 4
  Not Hispanic or Latino | 32 | 16 | 2 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 0 | 0 | 12
  White | 15 | 16 | 2 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 16 | 2 | 54

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival (PFS)
Description: PFS is the median amount of time subject survives without disease progression 6 months after treatment. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: At 6 months
Measure: Median (Full Range); unit: Months
Arm/Group | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) | Radiofrequency Ablation/Cryoablation (RFA/CA)
Number analyzed (Participants) | 36 | 1
Months | 2.8 [1.3 to 4.8] | NA [NA to NA] — Only one participant on the radiofrequency ablation/cryoablation group received the cryoablation, thus we cannot do the median on this group.

2. Secondary Outcome: Number of Grades 1-5 Adverse Events Related to Tremelimumab and Durvalumab
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v4.0. Grade 1 is mild, grade 2 is moderate, grade 3 is severe, grade 4 is life-threatening, and grade 5 is death related to adverse event.
Time Frame: 60 days after last treatment, an average of 44.89 months
Measure: Number; unit: adverse events
Arm/Group | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) | Radiofrequency Ablation/Cryoablation (RFA/CA)
Number analyzed (Participants) | 36 | 16
adverse events
  Grade 1 | 355 | 233
  Grade 2 | 125 | 133
  Grade 3 | 62 | 50
  Grade 4 | 6 | 3
  Grade 5 | 0 | 2

3. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 62 months and 3 days for the RFA/TACE group, and 27 months and 24 days for the RFA/CA group.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) | Radiofrequency Ablation/Cryoablation (RFA/CA)
Number analyzed (Participants) | 36 | 16
Participants | 36 | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 62 months and 3 days for the RFA/TACE group, and 27 months and 24 days for the RFA/CA group.
Arm/Group | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) | Radiofrequency Ablation/Cryoablation (RFA/CA)
All-Cause Mortality (participants affected / at risk) | 26/36 | 15/16
Serious Adverse Events (participants affected / at risk) | 20/36 | 7/16
Other Adverse Events (participants affected / at risk) | 36/36 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) (N=36) | Radiofrequency Ablation/Cryoablation (RFA/CA) (N=16)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, Skin rash near anus (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, Cellulitis - infection left upper extremity (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) (Infections and infestations) | 2 (2) | 0 (0)
Infections and infestations - Other, biliary stent infection (Infections and infestations) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Myasthenia Gravis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation/Trans-arterial Catheter Chemoembolization (RFA/TACE) (N=36) | Radiofrequency Ablation/Cryoablation (RFA/CA) (N=16)
Abdominal distension (Gastrointestinal disorders) | 4 (7) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 16 (24) | 7 (14)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 17 (32) | 7 (24)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 24 (65) | 13 (50)
Alkaline phosphatase increased (Investigations) | 26 (96) | 13 (42)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 32 (181) | 15 (55)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 31 (128) | 13 (52)
Autoimmune disorder (Immune system disorders) | 2 (3) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Bloating (Gastrointestinal disorders) | 11 (14) | 2 (3)
Blood and lymphatic system disorders - Other, aPTT decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 14 (60) | 9 (25)
Blurred vision (Eye disorders) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
CPK increased (Investigations) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (5) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (29) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Creatinine increased (Investigations) | 16 (76) | 6 (11)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 3 (5)
Dizziness (Nervous system disorders) | 4 (6) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 8 (9) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (10) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (13)
Edema limbs (General disorders) | 10 (15) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eye disorders - Other, Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Eye itching (Eye disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fatigue (General disorders) | 21 (36) | 12 (21)
Fever (General disorders) | 11 (13) | 9 (19)
Fibrinogen decreased (Investigations) | 3 (6) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Abdominal fullness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Epigastric pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, Chest soreness (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Muscle spasm (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Numbness - left hand (General disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (10) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 11 (18) | 7 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (47) | 5 (8)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (14) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 9 (18) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 6 (17) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 7 (43) | 3 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 28 (132) | 11 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (9) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (15) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 11 (32) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (20) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 30 (103) | 12 (25)
Hypophosphatemia (Metabolism and nutrition disorders) | 19 (53) | 6 (12)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (3) | 0 (0)
Immune system disorders - Other, Allergy development (Immune system disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, Skin rash near anus/groin (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, Headaches and nose bleeds (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Staph (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Thrush (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, cold sore (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8) | 4 (4)
Investigations - Other, Elevated TSH (Investigations) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 4 (4) | 0 (0)
Localized edema (General disorders) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 35 (243) | 13 (47)
Malaise (General disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Cramping - calves (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (18) | 8 (11)
Nervous system disorders - Other, Tongue numbness (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (35) | 1 (2)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 20 (36) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 25 (82) | 6 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (17) | 7 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (24) | 6 (8)
Respiratory failure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Pulmonary abnormalities (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, SOB (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 21 (130) | 3 (7)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Abrasion on forehead (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Brown lesion/rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Cracked skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Dermatitis - penis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Dermatitis - right buttocks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Face swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Itching (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Skin and subcutaneous tissue disorders - Other, Itching arm and chest (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Itchy back (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Keratosis; frontal scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Mild rash on shoulder and sparsely on back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Plaque rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Psoriasis; lower back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Psoriasis; trunk, bilateral extremities, and dorsal hand
Skin and subcutaneous tissue disorders - Other, Redness to radiation area (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Swelling - left leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Swollen feet and ankles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Wound to gluteal folds (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, itching-anus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, swelling- ankle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, swelling- feet/legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (13) | 6 (7)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 4 (4) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 19 (100) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT02821754/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort: Affected Patient Consent (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02821754/ICF_001.pdf
  • Informed Consent Form: Drug Only Consent (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02821754/ICF_002.pdf
  • Informed Consent Form: Drug and Ablative Therapy Consent (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02821754/ICF_003.pdf